CLINICAL TRIAL: NCT06513468
Title: The Value of Adding Group Education (DESMOND Method) to the Standard Primary Care Education Practices in Changing Glycemic Control and Self-care Practices in Adults With Type II Diabetes Mellitus: A Randomized Controlled Intervention Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Primary Health Care Corporation, Qatar (Other Government)
Responsible Party: Principal Investigator, Engy Salah Mohamed Abdelhamed, Consultant Family Medicine, Primary Health Care Corporation, Qatar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PHCCQatar
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes self management; DESMOND; effect of diabetes self management on glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: The enrolled study participants will be randomized to receive either the standard personal health care (routine diabetes health education services) or a standard group health education (DESMOND) session
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The standard health education of primary care . (Active Comparator): The first group will receive a standard health education for self-care practices done by attending two appointments in our clinics with the health education and dietitian in a personal session. The HA1C blood test together with completing a brief questionnaire form measuring the Diabetes Self-Care Activities during the past three months will be done after 3 and, 6 months will be done.
  Interventions: Other: Group education session by DESMOND Program
- The standard group health education (DESMOND) session (Experimental): The second group will attend a group health education using a standard DESMOND method (10-12 patients for each session lasting for 6 hours over one day by certified DESMOND educator in the conference room of the health center). The HA1C blood test together with completing a brief questionnaire form measuring the Diabetes Self-Care Activities during the past three months will be done after 3 and, 6 months will be done.
  Interventions: Other: Group education session by DESMOND Program

INTERVENTIONS:
Other: Group education session by DESMOND Program — is a validated structured education program for people with type 2 diabetes and their family members or carers (as appropriate)' This management approach was advised by the National Institute for Health and Care Excellence (NICE) in the UK since 2008. The program consists of a 6-hour face-to-face education session delivered by two trained educators over one day or two half-days to a group of 8-12 people with newly-diagnosed or ongoing type 2 diabetes. Annual reinforcement and review are part of the program , it is delivered as a business and usual in the secondary healthcare system of Qatar. The program is culturally adapted for Qatar considering beliefs and other health festivities.
  Other Names: The Diabetes Education and Self-Management for Ongoing and Newly Diagnosed with Type II diabetes

SUMMARY:
The goal of this clinical trial is to assess the outcome of delivering the health education in a group format using the DESMOND program compared to the standard health education in newly diagnosed adults with type 2 diabetes mellitus . The main questions it aims to answer is:

Does adding group education (DESMOND method) to the standard primary care education practices is effective in changing glycemic control and self-care practices in adults with Type II Diabetes Mellitus .

The enrolled study participants will be randomized to receive either the standard personal health care or group health education (DESMOND) session. questionnaire form measuring diabetes self-care will be administered at baseline together with measurement of HbA1C. These measurements will be repeated after 3 and 6 months of the intervention for both study groups.

DETAILED DESCRIPTION:
1. Objectives: This pilot, single primary healthcare center study is designed to assess the effect of delivering the group health education DESMOND program as an add-on to the standard health education in type 2 diabetic patients.
2. Design: This is an analytic randomized controlled intervention study for adult patients who are newly diagnosed type II Diabetes Mellitus. The enrolled study participants will be randomized to receive either the standard personal health care (routine diabetes health education services) or a standard group health education (DESMOND) session. A standard questionnaire form measuring diabetes self-care will be administered at baseline together with measurement of HbA1C. These measurements will be repeated after 3 and 6 months of the intervention for both study groups.
3. Setting :The Family Medicine clinics in Airport Health Center in Primary care, Qatar.
4. Participants: Newly diagnosed type II Diabetes Mellitus aged more than 18 years.
5. Intervention: A six-hour structured group education program to be delivered by one certified DESMOND health educator compared with the standard care.
6. Main outcome measures : Blood HbA1C % at baseline (before starting the diabetes management protocol of PHCC), after 3, and 6 months of follow up. In addition, the Diabetes self-management score (DSMQ) after 3 and 6 months of receiving both the standard personal health education sessions and the tested group education (DESMOND) method.

ELIGIBILITY:
Inclusion Criteria:

1. Adult more than 18 years, newly diagnosed Type II diabetes mellitus (within 4 - 6 weeks of diagnosis) attending the Airport Health Care Center.
2. Not yet receiving any form of standard health education in PHCC.

Exclusion Criteria:

1. Using diuretics or cancer therapy.
2. Had enduring mental health problem.
3. Participants in another research study.
4. Inability to communicate in Arabic or English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Blood HbA1C % | before starting the diabetes standard care , after 3, and 6 months of follow up for both arms
  before starting the diabetes standard care , after 3, and 6 months of follow up for both arms
The Diabetes self-management score using the (DSMQ) | before starting the diabetes standard care , after 3, and 6 months of follow up for both arms
  The Diabetes self-management score (DSMQ) at baseline , after 3 and 6 months of receiving both the standard personal health education sessions and the tested group education (DESMOND) method

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Care Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
we will keep participant name and other data confidential. it will be stored confidentially with the researcher only, and he may access to the data or specimens, for further research purpose in future.